CLINICAL TRIAL: NCT07063199
Title: A Single-arm, Open-label Clinical Study Evaluating the Safety and Efficacy of Daratumumab in Elderly Patients With Primary Immune Thrombocytopenia
Brief Title: Anti-CD38 Antibody Treating Elderly Patients With Primary Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025062
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Immune Thrombocytopenia; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Daratumumab) (Experimental): 30 enrolled subjects: once a week x 4 doses Daratumumab Injection
  Interventions: Drug: Daratumumab Injection

INTERVENTIONS:
Drug: Daratumumab Injection — This study adopts a prospective, single arm, open design method. Thirty subjects were enrolled in the study and were treated with CD38 monoclonal antibody (Daratumumab 16mg/kg/w) for 4 weeks.
  The first stage is the main research stage (d1-w4), which is the core treatment period. The subjects will receive intravenous infusion of 16mg/kg Daratumumab once a week for 4 weeks to observe the safety and efficacy during treatment.
  The second stage (w5-w24) is the stage of withdrawal from the visit, mainly to observe the safety and continuous efficacy of Daratumumab after treatment.

SUMMARY:
To evaluate the safety and efficacy of Anti-CD38 Antibody in the treatment of elderly patients with primary immune thrombocytopenia in patients who have failed multiple treatment.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Therefore, there is still a lack of effective treatment for adult ITP, especially for recurrent and refractory ITP patients, which is one of the problems that have attracted more attention and need to be solved urgently.The elderly are at a higher risk of developing immune thrombocytopenia, and they often have cardiovascular risk factors. They usually cannot tolerate treatment regimens such as hormones and immunosuppressants.

The main pathogenesis of ITP is the loss of platelet autoantigen immune tolerance, which leads to abnormal activation of humoral and cellular immunity. It is characterized by antibody mediated platelet destruction and insufficient platelet production by megakaryocytes. The residual long-term autoreactive plasma cells may be a source of therapeutic resistance to autoimmune cytopenia. Antiplatelet specific plasma cells have been detected in the spleen of patients with rituximab refractory ITP. Therefore, the strategy of simply eliminating B cells may not work, because LLPC will continue to produce pathogenic antibodies. However, targeting LLPC becomes a new strategy to treat autoimmune diseases.

Daratumumab, a kind of anti-CD38 antibody, is a new type of monoclonal antibody targeting CD38. It targets plasma cells and has carried out some clinical studies in multiple myeloma, with good therapeutic effects. In addition, the clinical trials of daratumumab in the treatment of autoimmune diseases, including membranous nephropathy, systemic lupus erythematosus (SLE) and ITP, are also being carried out simultaneously. The investigators assume that autologous reaction LLPC may be the cause of treatment failure in some ITP patients. Therefore, the use of CD38 monoclonal antibody to clear long-term surviving plasma cells in ITP patients may be a new strategy for treating ITP patients.Our hospital has conducted and completed a clinical trial of daratumumab for the treatment of adult ITP. The dosage was 16mg/kg/w for a total of 8 weeks. The results showed that for refractory patients who had previously received multiple lines of treatment with poor efficacy, daratumumab could rapidly increase platelet counts. The median onset time was about 1 week. At 24 weeks of follow-up, the effective rate was approximately 60%, and no serious adverse events occurred. The efficacy and safety were confirmed, but the number of elderly patients included was relatively small.

Therefore, the investigators designed this clinical trial to evaluate the safety and efficacy of daratumumab in the treatment of elderly patients with immune thrombocytopenia in patients who failed multiple treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years, male or female.
* Before enrollment, the subjects have been clinically diagnosed with primary immune thrombocytopenia for no less than three months according to the American Society of Hematology guidelines 2011 Evidence-Based Practice Guideline (Neunert et al. 2011) or the International Consensus Report for the Investigation and Management of Primary Immune Thrombocytopenia (Provan et al. 2010), as applicable locally.
* Patients have failed glucocorticoid therapy and at least one standard second-line therapy. (either due to inefficacy, efficacy could not be maintained, or relapse). Patients should have a history of response to previous ITP standard first-line therapy (glucocorticoids and/or intravenous human immunoglobulin) (PLT≥50×10^9/L);
* Platelet count <30×10^9/L within 24 hours before the first administration of the study drug; During the screening period, platelet counts were measured at least 2 times (at least 1 week apart), with an average platelet count <30×10^9/L and no platelet count > 35×10^9/L.
* ECOG performance status score of ≤2.
* Enrollment of subjects receiving maintenance therapy is permitted, including glucocorticoids (≤0.5 mg/kg of prednisone or equivalent) or TPO receptor agonists. Only one concomitant medication was allowed at the time of enrollment, and the concomitant medication must have been stable for a minimum of 4 weeks prior to the first dose of the study drug.
* For fertile female patients, a negative pregnancy test result is required. Fertile female and male patients must use effective contraception separately during the study and for 4/6 months after the cessation of study drug treatment.
* Subjects comprehensively understand and can adhere to the study protocol requirements and willingly signed the informed consent form.

Exclusion Criteria:

* Those who are allergic to anti-CD38 monoclonal antibody or excipients, or who have received anti-CD38 monoclonal antibody in the past and failed or kept a continuous response of less than 6 months.
* All kinds of secondary thrombocytopenia or autoimmune hemolytic anemia.
* Any history of thrombotic or embolic events or extensive and severe bleeding, such as hemoptysis, massive upper digestive tract hemorrhage, intracranial hemorrhage, etc., or sepsis or other irregular bleeding within 12 months before the first medication.
* Participated in or was exposed to any other investigational drug study (including vaccine study) during the 4 weeks or 5 half-lives (whichever is older) prior to the first dose.
* Subjects taking antiplatelet drugs within 3 weeks before the first dose.
* Subjects who have received emergency treatment for ITP (e.g., methylprednisolone, platelet transfusion, intravenous immunoglobulin infusion, or thrombopoietin receptor agonist therapy) within 2 weeks prior to the first dose of study drug.
* Subjects who have been treated with medications including azathioprine, danazol, dapsone, cyclosporine A, tacrolimus, and sirolimus within 4 weeks prior to the first dose of study drug. Subjects who have receive anti-CD20 monoclonal antibodies such as rituximab, or medications including cyclophosphamide and vindesine within 6 months prior to the first dose of study drug.
* Subjects who have undergone splenectomy within 6 months prior to the first dose of study drug.
* Subjects who have received live vaccines within 4 weeks prior to the first dose of study drug, or plan to receive any live vaccines during the course of the study.

Subjects who are diagnosed with Myelodysplastic syndromes (MDS); Subjects with a with a history of malignancy within the 5 years prior to screening (excluding completely cured in situ cervical cancer and non-metastatic skin squamous cell carcinoma or basal cell carcinoma).

* Subjects who have undergone allogeneic stem cell transplantation or organ transplantation.
* Subjects with a clinically significant medical history, as perceived by investigators, that will pose risks to subjects' safety during the study or potentially affect the safety or efficacy analyses, includes major clinical histories such as circulatory system abnormalities, endocrine system abnormalities, nervous system diseases, blood system diseases, immune system diseases, mental diseases and metabolic abnormalities and so on. e.g., subjects with acute myocardial infarction, unstable angina pectoris, or severe arrhythmias (multifocal ventricular premature contractions, ventricular tachycardia, or ventricular fibrillation) within the 6 months before screening ; New York Heart Association (NYHA) class III-IV heart failure; subjects who were known to have had moderate or severe persistent asthma or chronic obstructive pulmonary disease within the 5 years prior to screening, or whose condition was currently poorly controlled;
* Subjects with a history of severe recurrent or chronic infections, or acute infections requiring systemic treatment with antibiotics, antiviral drugs, antiparasitic drugs, anti-amoebic drugs, or antifungal drugs within 4 weeks prior to the first dose and during the screening period, or superficial skin infections requiring systemic treatment within one week prior to the first dose of study drug. Notably, after the resolution of the infection, the subject may be re-screened.
* Subjects with a history of known or suspected immunosuppression, including invasive opportunistic infections such as histoplasmosis, listeriosis, coccidioidomycosis, pneumocystis pneumonia, and aspergillosis, even if the infection has resolved; or unusually frequent, recurrent, or prolonged infections (as judged by the investigator).
* Significant laboratory abnormalities during screening included:

  1. Alanine aminotransferase or aspartate aminotransferase greater than three times the upper limit of normal (ULN).
  2. Total bilirubin greater than 1.5 times the ULN (note: subjects diagnosed with Gilbert syndrome based on medical records should not be excluded based on this criterion).
  3. absolute neutrophil count < 1500/mm3.
  4. hemoglobin < 9g/dL; IgG < 500 mg/dL.
  5. lymphocyte count < 500/mm3.
  6. Creatinine clearance (CrCl) < 30 mL/min (i.e., CrCl ≥30 mL/min is allowed)
* Positive for HIV antibodies or syphilis antibodies.
* Subjects test positive for Hepatitis B surface antigen (HBsAg) or subjects test positive for hepatitis B core antibody and HBV-DNA (through polymerase chain reaction testing), or subjects test positive for hepatitis C virus antibody and HCV-RNA during the screening period. Subjects with positive hepatitis B core antibody but negative HBV-DNA can be enrolled, with HBV-DNA monitoring every 4 weeks.
* Pregnant or lactating women, or those intending to conceive or breastfeed during the study; and male partners intending to induce pregnancy during the study.
* Any other conditions unsuitable for participation in this study, as assessed by the investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events of Anti-CD38 antibody treatment | 24 weeks
  Incidence, severity, and relationship of treatment emergent adverse events after Anti-CD38 antibody treatment
Efficacy after Daratumumab treatment within 8 weeks | 8 weeks
  Evaluation of ORR (overall response rate) within 8 weeks after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RAs or corticosteroids during the study period

SECONDARY OUTCOMES:
CR (complete remission) ratios at each visit time point | 24 weeks
  Evaluation of CR（complete remission) ratios at each visit time point after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RAs or corticosteroids during the study period
ORR (overall response rate) at each visit time point | 24 weeks
  Evaluation of ORR (overall response rate) at each visit time point after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RAs or corticosteroids during the study period
Other efficacy evaluation | 24 weeks
  Proportion of subjects achieving platelet counts ≥ 50×10^9/L at least once in absence of rescue therapy, and without having had dose increment of TPO-RAs or corticosteroids at each visit time poin
Time to response (TTR) | 24 weeks
  Duration from treatment initiation to platelet count ≥30×10^9/L and at least twice the baseline without having received any platelet elevating therapy or having had dose increment of TPO-RAs and/or corticosteroids
Sustained response time-1 | 24 weeks
  The cumulative time of platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count during the study period.
Sustained response time-2 | 24 weeks
  The cumulative time of platelet count ≥ 50 × 10^9/L during the study period.
Emergency treatment | 24 weeks
  Percentage of patients who need emergency treatment during the study period.
Reduction of concomitant drug after anti-CD38 antibody treatment by week 12 | 12 weeks
  Percentage of patients with reduced doses of corticosteroids and/or other concomitant immunosuppressive drugs at baseline by 12 weeks of anti-CD38 antibody treatment
Number of subjects with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale | 12 weeks
  Changes of the subjects' numbers in WHO bleeding score after anti-CD38 monoclonal antibody treatment according to the reported World Health Organization's Bleeding Scale at week 12. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital; Yunfei Chen, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months to 36 months after study completion.
Supporting Information: SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI